CLINICAL TRIAL: NCT02582463
Title: Development of the Medicines Optimisation Assessment Tool (MOAT) - Targeting Hospital Pharmacists' Input to Reduce Risks and Improve Patient Outcomes
Brief Title: Development of the Medicines Optimisation Assessment Tool
Acronym: MOAT
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 15/0525; CDRF-2014-05-033 (Other Grant/Funding Number: National Institute for Health Research (NIHR))
Record Dates: First submitted 2015-10-12; First posted 2015-10-21 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2017-10

CONDITIONS: Medicines Optimisation
Keywords: Risk Assessment; Hospitals; Pharmacists; Medication Systems; Patient Selection; Prognosis research

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop a prediction-tool, the Medicines Optimisation Assessment Tool (MOAT), to assist hospital pharmacists identify patients at highest risk of preventable medication related problems (MRPs). This has the potential to permit pharmacists to identify and focus on the small number of patients (approximately 6%) who are likely to experience a significant MRP while in hospital.

DETAILED DESCRIPTION:
The purpose of this study is to develop a prediction-tool, the Medicines Optimisation Assessment Tool (MOAT), to assist hospital pharmacists identify patients at highest risk of preventable medication related problems (MRPs).

The MOAT will be developed following recommendations of the PROGnosis RESearch Strategy (PROGRESS) partnership. A prospective cohort study of 1,500 patients will be used to develop the MOAT from the medical wards of two UK hospitals. Data will be collected on prognostic factors (selected based on a review of published literature and expert opinion) for each patient, together with details of MRPs that occur. All MRPs will be reviewed by an expert panel who will grade for severity and preventability using recognised criteria. Multivariable logistic regression models will be used to determine the relationship between potential risk factors such as polypharmacy, renal impairment, and the use of 'high risk' medicines, and the study outcome of preventable medication related problems that are at least moderate in severity. Bootstrapping will be used to adjust the MOAT for optimism, and predictive performance will be assessed using calibration and discrimination. A simplified scoring system will also be developed, which will be assessed for sensitivity and specificity.

The intention of this research is to develop a prediction-tool (the MOAT), which has the potential to be adopted widely into clinical practice. If the initial research is successful in producing a prediction-tool with good predictive performance further research will be carried out to assess how feasible it would be to use the MOAT in practice, the potential efficiency savings, and an assessment of clinical risk to patients through use of the MOAT.

ELIGIBILITY:
Inclusion Criteria:

* subject admitted to the Medical Division (General, Emergency, and Elderly Medicine) at the study sites

Exclusion Criteria:

* subject admitted for investigation-only
* subject not prescribed medication
* subject both admitted and subsequently discharged outside of core pharmacy working hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Medical Division (General, Emergency, and Elderly Medicine) at the Luton and Dunstable University Hospital and Watford General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1552 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Number of MRPs experienced by study participants | Through study completion (discharge from hospital), an average of 6 days
  The outcome measure (i.e. all MRPs) will be graded for severity and preventability, then multivariate analysis such as logistic regression models will be used to determine the relationship between predictors (prognostic factors) and the outcome (MRPs which are at least moderate in severity and preventable). The objective will be to find the best combinations of predictors that are highly sensitive for detecting the outcome measure while achieving the maximum possible specificity.

SECONDARY OUTCOMES:
Feasibility of using the MOAT (content validity and ease of use) | 18 months
  Content validity will be assessed to ensure that clinicians consider the items in the MOAT to be clinically sensible, no obvious items are missing, the method of grouping the individual predictors is reasonable, and the items seem appropriate for the purpose of the tool. Ease of use depends on the length of time needed to apply the tool and the simplicity of interpretation. A consensus development technique will be used to generate consensus on content validity and simplicity of interpretation. Time to apply the MOAT will be assessed by observation.
Potential efficiency savings | 18 months
  The impact of the MOAT in terms of potential workload for pharmacists will be informed by the number of patients who screen positive (from internal validation). This will indicate the proportion of patients who would be expected to require review by a pharmacist, i.e. the total number that pharmacists would need to see to identify those at highest risk of MRPs.
Potential clinical risk to patients through use of the MOAT | 18 months
  Patients who experience an MRP but would be excluded from pharmacist review by the MOAT (i.e. false negatives) will be reviewed in detail to identify the potential clinical risk (i.e. severity of missed events).

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Geeson, Principal Investigator — University College, London
Locations (1):
- Luton and Dunstable University Hospital, Luton, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geeson C, Wei L, Franklin BD. Medicines Optimisation Assessment Tool (MOAT): a prognostic model to target hospital pharmacists' input to improve patient outcomes. Protocol for an observational study. BMJ Open. 2017 Jun 14;7(6):e017509. doi: 10.1136/bmjopen-2017-017509. PMID 28615279